CLINICAL TRIAL: NCT05345834
Title: Advancing Perinatal Mental Health and Well-Being: The DC Mother-Infant Behavioral Wellness Program
Brief Title: The DC Mother-Infant Behavioral Wellness Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: George Washington University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Catherine Limperopoulos, Director of the Developing Brain Institute and Director of the Advanced Pediatric Brain Imaging Research Program, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00015379
Record Dates: First submitted 2022-03-02; First posted 2022-04-26 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Perinatal Depression; Perinatal Anxiety; Prenatal Stress
Keywords: Postpartum depression; postpartum anxiety; pregnancy; Black women; stress; Anxiety; Depression
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders; Depression | interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: Women in the patient navigator arm (Group 2a) can choose to participate in group-based preventive interventions based on: (1) a culturally adapted CBT (in person within prenatal care site or virtual given COVID); (2) peer support group (virtual); or (3) both. Women in the threshold risk group (Group 2b) at baseline warrant treatment interventions and will be invited to participate in: (1) culturally adapted CBT (individual, in person or virtual given COVID); (2) peer support (virtual); or (3) both. Women in this more severe risk group may be referred for psychiatric treatment if warranted. Randomization lists will be generated by the study statistician using a permuted block design and uploaded to a HIPAA-compliant, password-protected website (REDCap) allowing for patient randomization at the time of registration in the data collection system.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants will participate in usual prenatal care throughout the duration of study.
- Patient Navigation and treatment (Experimental): In the patient navigation arm, women who do not meet diagnostic criteria (Group 2a) can participate in: (1) group-based CBT preventative intervention; (2) peer support group (virtual); or (3) both. Women in the threshold risk group, meeting diagnostic criteria for depression/anxiety (Group 2b) at baseline can participate in: (1) individual CBT treatment (2) peer support group (virtual) (3) both
  Prevention group includes 8 sessions based on culturally adapted CBT for Black/ of African descent populations facilitated by mental health professionals. Individual treatment includes 12 sessions based on culturally adapted CBT for Black/ of African descent populations.
  Interventions: Behavioral: Patient Navigation; Behavioral: Adapted Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: Patient Navigation — Participants in arm 2 will receive patient navigation provided by humans (rather than e-navigation) to provide personalized care to include support, resources, and referrals to address psychosocial issues that arise during the perinatal period. Patient navigation is available to participants through 12 months postpartum.
  Other Names: Maternity Care Specialist
  Arms: Patient Navigation and treatment
Behavioral: Adapted Cognitive-Behavioral Therapy — Participants who do not meet diagnostic criteria (Group 2a) will participate in a prevention group which includes 8 sessions based on culturally adapted CBT for Black/ of African descent populations facilitated by mental health professionals. Participants who meet diagnostic criteria (Group 2b) will participate in individual treatment which includes 12 sessions based on culturally adapted CBT for Black/ of African descent populations.
  Other Names: Adapted CBT
  Arms: Patient Navigation and treatment

SUMMARY:
This randomized controlled study will examine the effectiveness of patient navigation with culturally adapted cognitive-behavioral interventions and peer support groups for low-income Black/of African Descent pregnant women who are experiencing stress, anxiety, and/or depression.

DETAILED DESCRIPTION:
The overarching objective is to develop and evaluate a collaborative, multi-dimensional and culturally tailored community-based model of integrated perinatal MH care. The target population is low-income Black/of African descent women with pregnancy-related stress, anxiety, and depression. There are two specific aims: (1) to refine an individualized plan to integrate patient navigation and a culturally adapted cognitive-behavioral (CBT) intervention for low-income Black/of African Descent women designed to increase recruitment and retention within the healthcare community system, and (2) through a two-arm prospective randomized controlled design, women who are subthreshold and threshold risk for prenatal stress, depression and/or anxiety will participate in one of two interventions: (a) existing prenatal intervention (usual care); or (b) patient navigation plus culturally adapted CBT, and peer support groups.

The investigators will screen 1,000 low-income pregnant AA women (18-45 years of age) in their second pregnancy visit with validated tools for stress, anxiety, and depression. A total of 700 study participants will be recruited from urban prenatal care centers in the Washington DC area and will be randomized Usual Care of Intervention conditions above (n=350/condition). Following randomization, participants will participate in a diagnostic interview based on DSM-5 criteria to 'self-select' themselves into 1 of 2 groups (i.e., 'threshold' or 'subthreshold'). Threshold includes women who meet criteria for depression or anxiety based on DSM-5 diagnostic criteria. Subthreshold includes all other women who do not meet DSM criteria). In the intervention arm, participants in the threshold group will receive a 1:1 CBT treatment intervention, and participants in the subthreshold group will receive a group CBT intervention. Both threshold groups will also include patient navigation and participation in a peer support group. Participants will complete standardized health, mental health, and well-being questionnaires during pregnancy at their prenatal site, and up to 12 months after delivery at their well-baby visits, when they also will complete questionnaires about their infants' development and behavior. All infants also will undergo a standardized developmental test at 12 months. Health care utilization and outcomes also will be collected through electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Black/of African Descent
* Pregnant (gestational weeks ≤ 28 weeks)
* Age 18-45
* English proficient
* Receiving services in 1 of 4 study sites above
* Low-income: i.e., receiving Medicaid
* Subthreshold or threshold risk for maternal distress (stress, depression, and/or anxiety)
* Able to provide consent

Exclusion Criteria:

* age <18
* Currently under the influence of a substance(s)
* Experiencing psychosis
* Critical (clinical) risk: actively suicidal or homicidal
* Not Black/of African Descent
* Planning to deliver outside DC

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 700 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Stress at 24 weeks of pregnancy to 12 months postpartum | Stress will be measured at 24 weeks of pregnancy through infant age of 12 months
  Perceived Stress Scale: A 10-item questionnaire to measure the self-reported level of stress in the respondents by assessing feelings and thoughts during the last month. Each item is scored from 0 (never) to 5 (very often) with a range of 0 to 40 for the total score of the scale. A higher level of stress is indicated by higher scores on this scale.
Change in Depression at 24 weeks of pregnancy to 12 months postpartum | 2nd Obstetrics visit (assessed 24-28 weeks gestation) through 12 months postpartum
  Edinburgh Postnatal Depression Scale: A 10-item scale used to indicate whether a parent has symptoms that are common in women with depression during pregnancy and in the year following the birth of a child. Each item is scored from 0 (As much as I ever did) to 3 (Not at all) with a range of 0 to 30. Higher level of depression is indicated by a higher score on this scale.
Change in Anxiety at 24 weeks of pregnancy to 12 months postpartum | 2nd Obstetrics visit (assessed 24-28 weeks gestation) through 12 months postpartum
  General Anxiety Disorder-7 (GAD-7): A 7-item scale to measure levels of anxiety in respondents by assessing feelings and thoughts over the past 2 weeks. Each item is scored from 0 (Not at all) to 3 (Nearly every day) with a range of 0 to 21. Higher level of depression is indicated by a higher score on this scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Unity Healthcare - Brentwood, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Le HN, Andescavage N, Keller JM, Bassa MM, Danielson AL, Henderson D, Bond S, Mjenga N, Wells S, Quinn P, Limperopoulos C. Protocol for a randomized controlled trial of the Mommy&Me study: A multi-modal approach to address social determinants of health and mental health among low-income Black perinatal populations. Contemp Clin Trials Commun. 2025 Apr 21;45:101489. doi: 10.1016/j.conctc.2025.101489. eCollection 2025 Jun. PMID 40336702

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT05345834/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT05345834/ICF_001.pdf